CLINICAL TRIAL: NCT04015115
Title: Youth Opioid Recovery Support (YORS): Improving Care Systems for Young Adults With Opioid Use Disorder
Brief Title: Youth Opioid Recovery Support: Improving Care Systems
Acronym: YORS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Victoria Selby, Assistant Professor, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-0085682
Record Dates: First submitted 2019-07-01; First posted 2019-07-10 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-01

CONDITIONS: Opioid-Related Disorders
Keywords: Buprenorphine; Central Nervous System Depressants; Chemically-Induced Disorders; Community Mental Health Services; Drug Partial Agonism; Heroin Dependence; Medication Adherence; Mental Disorders; Naltrexone; Narcotic Antagonists; Narcotics; Opioid-Related Disorders; Opioid Substitution Treatment; Patient Compliance
MeSH Terms: conditions — Opioid-Related Disorders; Chemically-Induced Disorders; Heroin Dependence; Medication Adherence; Mental Disorders; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Youth Opioid Recovery Support service model (Experimental): The components of the Youth Opioid Recovery Support service model includes 1) home-delivery of standard-of-care medication and individual/family counseling services; 2) assertive outreach efforts by the treatment team; and 3) contingency management incentives upon receipt of medication treatment.
  Interventions: Behavioral: Youth Opioid Recovery Support service model

INTERVENTIONS:
Behavioral: Youth Opioid Recovery Support service model — see arm 1 description

SUMMARY:
Opioid addiction, also referred to as opioid use disorder, among young people is a growing health concern for patients and their families. Overdose deaths related to opioids have been steadily increasing in number and are at an all-time high. Opioid addiction has serious consequences such as getting HIV, legal problems, relationship problems, and unemployment.

Currently, there are two standard of care office-based medications available to treat opioid use disorder, buprenorphine and naltrexone. Naltrexone has been available for several years as an extended-release monthly injectable formulation, and more recently buprenorphine is as well. Both of these medications are typically administered in the medical office setting. Long-acting injection medications like these help people that may otherwise forget doses, skip doses, and relapse.

MAT that are FDA-approved such as these paired with counseling can help sustain recovery, but retention to treatment is a concern, especially among young adults. Many barriers arise for attending office-based treatment (e.g., transportation) often resulting in falling away from treatment and relapsing. Involvement of family members is often challenged by health care provider concerns about patient privacy, and existing relationship strain between patients and their families.

The Youth Opioid Recovery Support (YORS) treatment delivery model hopes to address barriers to retention to substance treatment among those with opioid use disorder who have already decided to get treatment with either extended-release naltrexone or extended-release buprenorphine. The YORS model involves: 1) home-delivery of standard-of-care medication and individual/family counseling services; 2) assertive outreach efforts by the treatment team; and 3) contingency management incentives upon receipt of treatment.

This service model has already shown promise in addressing barriers to treatment retention particularly difficulties with medication adherence in patients who were prescribed monthly injectable extended-release naltrexone. Now that extended-release buprenorphine is also available, broader MAT options provided in an assertive service delivery model may maximize treatment retention and recovery outcomes. Further, transitioning participants from home-based receipt of treatment to clinic-based care begins the translation to sustainable health care.

ELIGIBILITY:
Inclusion Criteria:

* Young adults, ages 18-26, admitted to residential/inpatient addiction treatment
* Meets DSM-5 criteria for opioid use disorder
* Has used opioids other than specifically prescribed within 30 days prior to consent
* Has selected treatment with extended-release naltrexone or extended-release buprenorphine
* Is prescribed extended-release naltrexone or extended-release buprenorphine under the care of a Mountain Manor Treatment Center physician or nurse practitioner
* Willing to designate one or more family members of their choice to be involved with their treatment.
* Family Participant: must be at least 18 years old, be designated by the patient Participant, and willing to be involved in the treatment.

Exclusion Criteria:

* Living situation is beyond a reasonable travel distance from the treatment center
* Currently, in jail, prison, or any inpatient overnight facility as required by course of law or have a pending legal action which may prevent an individual from completing the study

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2019-07-26 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Retention in medication-assisted treatment of opioid use disorder | Measured every 4 weeks for the duration of enrollment, up to 36 weeks, by examining participants medical record.
  Total number of outpatient doses of extended-release naltrexone or extended-release buprenorphine received by the participant between enrollment and the end of the study window
Opioid relapse | Self report and urine specimens will be collected every 2 weeks for the duration of enrollment, up to 36 weeks.
  Opioid Relapse is defined as 10 days of opioid use within a 28-day period. Days of opioid use are calculated using data from self report and urine toxicology with missing or positive urine specimens imputed as 5 days of use.
Total number of opioid positive drug screens | Every 2 weeks for the duration of enrollment, up to 36 weeks.
  Urine drug screening will objectively determine opioid use or nonuse.

SECONDARY OUTCOMES:
Change in behaviors related to recovery | Participants will be assessed at baseline (time of enrollment into the study), then, every 4 weeks, up to 36 weeks.
  Participant-reported behaviors associated with function (e.g., employment), legal involvement, HIV risk behavior, overdoses, and crisis utilization (emergency room visit, hospitalization, detoxification services).
Continued receipt of care post-intervention | Continued care will be assessed at one time-point 1 month following the YORS intervention period of the study.
  Receipt of medication-assisted treatment at the treatment center after the last dose of home-delivered medication.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Fishman, MD, Principal Investigator — Mountain Manor Treatment Center; Kevin Wenzel, PhD, Study Director — Mountain Manor Treatment Center; Victoria Selby, PhD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- Mountain Manor Treatment Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No